CLINICAL TRIAL: NCT04386967
Title: Open and Incremental Phase I Clinical Trial of Recombinant Human GM-CSF Type II Herpes Simplex Virus (OH2) Injection (Vero Cells) in the Treatment of Advanced Solid Tumors
Brief Title: OH2 Injection in Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Binhui Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OH2-I-ST-01
Record Dates: First submitted 2020-04-13; First posted 2020-05-13 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor; Melanoma
Keywords: Oncolytic Virus
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose expansion (Experimental): Dose expansion trial comprises of 2 cohorts. In cohort 1, OH2 injection will be administered at 1x10e7CCID50/mL . In cohort 2, OH2 injection will be administered at 1x10e7CCID50/mL in combination with Keytruda injection, an anti-PD-1 antibody, and the first doses of the two anti-tumor agents will be administered on the same day.
  Interventions: Biological: OH2 injection; Drug: Keytruda

INTERVENTIONS:
Biological: OH2 injection — Oncolytic Type 2 Herpes Simplex Virus
Drug: Keytruda — Anti-PD-1 antibody
  Other Names: pembrolizumab

SUMMARY:
This phase I study evaluates the safety and efficacy of OH2 as single agent or in combination with Keytruda, an anti-PD-1 antibody, in patients with malignant solid tumors (Melanoma).

OH2 is an oncolytic virus developed upon genetic modifications of the herpes simplex virus type 2 strain HG52, allowing the virus to selectively replicate in tumors. Meanwhile, the delivery of the gene encoding human granulocyte macrophage colony-stimulating factor (GM-CSF) may induce a more potent antitumor immune response.

ELIGIBILITY:
Inclusion Criteria:

1. The non-operative stage III or stage IV malignant tumor patients with clear diagnosis by pathology and/ or cytology; breast cancer, gastrointestinal adenocarcinoma, liver cancer, cervical cancer, malignant melanoma, head and neck tumors, Priority inclusion in soft tissue sarcomas (mainly for melanoma patients at the dose extension phase).
2. The absence of a conventional effective treatment or treatment failure or recurrence by a conventional method.
3. Male or female patients, aged 18 ≤ 75 years (including boundary value), general physical condition score ECOG 0 ≤ 1, expected survival time more than 3 months.
4. Prior anti-tumor treatment (including endocrine, chemical/ radiotherapy,targeted therapy) was over 4 weeks (more than 6 weeks of discontinuation using nitroso-and mitomycin-based chemotherapy) and was recovered to grade 1 from the side effects of prior treatment.
5. Those who have undergone major surgery will have to undergo surgery for four weeks.
6. There is at least one measurable lesion that is suitable for intratumoral injection. According to RECIST version 1.1, it is determined that at least once the CT or MRI examination shows the tumor lesion, it is possible to measure the tumor focus. The measured tumor focus is defined as the longest diameter ≥ 10 mm and the scanning thickness is not more than 5.0 mm. For lymph node lesions, the short diameter is ≥ 15 mm.
7. There is no serious dysfunction of the main organs.
8. (a) WBC≥3.0×109／L，ANC≥2.0×109／L ，PLT≥100×109／L，Hb≥90 g/L； (b) BUN and Scr. were in the upper limit of 1.5 times of the normal value; (c) TBIL≤ 1.5 times the upper limit of the normal value. (d) ALT and AST ≤ 2.5 times the upper limit of normal value; The value of patients with liver metastasis did not exceed 5 times the upper limit of normal value. (e) Coagulation function is normal (PT and APPT are within 1.5 times of the upper limit of normal value).
9. Female subjects and their spouses received effective contraceptives during and within 3 months of treatment.
10. Subjects with herpes in the reproductive organs needed three months after the end of herpes.
11. The informed consent was voluntarily signed and the expected compliance was good.

Exclusion Criteria:

1. Severe medical diseases, including severe heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, severe infection, active digestive tract ulcer, abnormal immune function (including, but not limited to, rheumatoid arthritis, lupus erythematosus, Sjogren's syndrome, etc.).
2. History of primary grape-film melanoma or other malignant tumors in the 3 years prior to treatment. (use of combination drugs only)
3. Past or present immunodeficiency diseases. (use of combination drugs only)
4. Treated with PD-1/PD-L1 or PD-L2 monoantigens or inhibitors that have been used or used in the past. (use of combination drugs only)
5. Autoimmune diseases requiring systemic treatment (e.g. steroids or immunosuppressants) during the first 2 years of treatment, such as autoimmune pneumonia, glomerular nephritis, vasculitis and other symptoms of autoimmune diseases; Except for wind or child asthma. (use of combination drugs only)
6. Have uncontrolled primary or brain metastatic tumors.
7. Suffering from uncontrolled mental illness, infectious diseases.
8. The lesions cannot meet the requirements of injection capacity in the tumor body.
9. Pregnant or lactating women.
10. Other experimental therapies or antiviral therapy are used or are being used within 4 weeks of treatment.
11. Other clinical studies have been taken in the past 4 weeks.
12. Allergy to herpes virus and drug ingredients.
13. The researchers believe that there is any reason why the patient is not suitable to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-22 (Actual); Primary Completion 2026-03-13 (Estimated); Study Completion 2026-12-13 (Estimated)

PRIMARY OUTCOMES:
Further evaluation of dose-limiting toxicity (DLT) and maximum-tolerated dose (MTD) of OH2 in patients with solid tumors | 12 months
The dose-limiting toxicity (DLT) of OH2 injection and Keytruda in patients with solid tumors | 12 months
The maximum-tolerated dose (MTD) of OH2 injection in combination with Keytruda in patients with solid tumors | 12 months

SECONDARY OUTCOMES:
The response rate of patients with solid tumors receiving OH2 injection monotherapy and OH2 injection in combination with Keytruda | 12 months
The biodistribution of OH2 injection as determined by the concentration of OH2 in blood, urine and feces of participating patients | 12 months
The immunogenicity of OH2 injection as determined by the detection of antibodies in response to OH2 and GM-CSF | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang X, Tian H, Chi Z, Si L, Sheng X, Hu H, Gu X, Li S, Li C, Lian B, Zhou L, Mao L, Tang B, Yan X, Wei X, Li J, Liu B, Guo J, Kong Y, Cui C. Oncolytic virus OH2 extends survival in patients with PD-1 pretreated melanoma: phase Ia/Ib trial results and biomarker insights. J Immunother Cancer. 2025 Feb 6;13(2):e010662. doi: 10.1136/jitc-2024-010662. PMID 39915002